CLINICAL TRIAL: NCT00529724
Title: Mechanisms of Body Weight Gain in Patients With Parkinson's Disease After Subthalamic Stimulation
Brief Title: Body Weight Gain, Parkinson, Subthalamic Stimulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Franck Durif, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHU-0024
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Parkinson's Disease
Keywords: Energy metabolism, metabolic syndrome, by chronic bilateral subthalamic stimulation, Parkinson's disease; Patients with Parkinson's disease and will be treated by chronic bilateral subthalamic stimulation.
MeSH Terms: conditions — Parkinson Disease; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Energy metabolism by chronic bilateral subthalamic stimulation — Patients will be studied before and after STN-DBS surgery

SUMMARY:
Chronic bilateral subthalamic stimulation leads a spectacular clinical improvement in patients with motor complications. However, the post-operative body weight gain involved may limit the benefits of surgery and induce critical metabolic disorder. The aim of this study to determine the energy expenditure in usual conditions of life.

DETAILED DESCRIPTION:
Patients will be studied before (between 3 and 1 months) and after (1 month) STN-DBS surgery. Each time the same measurements will be taken. The principal ones will be :

* Clinical examination
* Autoevaluation dietary questionnaire
* Biological tests
* Study in calorimetry chamber (only in Clermont-Ferrand centre)
* Heart rate recorded during 7 days in usual conditions of life
* Energy expenditure recorded during 14 days in usual conditions of life with normalized water (18O 10 %) and Deuterium oxide (99.94 %D)
* Acute Ldopa challenge (in both conditions of dopa and stim)
* Apathy evaluation
* Body weight, and body compositions measurements

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years old
* Diagnosis of Parkinson' disease established for 5 years at least
* Ldopa effect > 50 %
* Hoehn and Yarh score > 2.5 in On phase

Exclusion Criteria:

* Metabolism disorder
* Biological analysis abnormal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-09-03 (Actual); Primary Completion 2015-09-21 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
heart rate recorded during 7 days in usual conditions of life | 7 days in usual conditions of life
energy expenditure recorded during 14 days in usual conditions of life with normalized water (18O 10 %) and Deuterium oxide (99.94 %D) | 14 days in usual conditions of life

CONTACTS AND LOCATIONS:
Overall Officials: Franck Durif, Pr, Principal Investigator
Locations (1):
- CHU, Clermont-Ferrand, France